CLINICAL TRIAL: NCT03945487
Title: Safety and Efficacy of Human Unbilical Cord Derived-mesenchymal Stem Cells Treatment for Patients With Decompensated Liver Cirrhosis
Brief Title: Mesenchymal Stem Cells Treatment for Decompensated Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Treatment and Research Center for Infectious Diseases, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-011
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Decompensated Liver Cirrhosis
Keywords: liver cirrhosis; mesenchymal stem cells; safety; liver function
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive treatment plus UC-MSC treatment (Experimental)
  Interventions: Biological: umbilical cord-derived mesenchymal stem cell
- Comprehensive treatment (Other)
  Interventions: Other: Comprehensive treatment

INTERVENTIONS:
Biological: umbilical cord-derived mesenchymal stem cell — Taken a dose of 1.0*10E6 UC-MSC/kg body weight intravenously three times at 3-week intervals, in addition to comprehensive treatment.
  Arms: Comprehensive treatment plus UC-MSC treatment
Other: Comprehensive treatment — 1. All patients received anti-HBV treatment with NAs (entecavir (ETV), tenofovir disoproxil fumarate (TDF), or tenofovir alafenamide (TAF)).
  2. Strategies based on targeting abnormalities in gut-liver axis by antibiotic administration (i.e. rifaximin), improving the disturbed systemic circulatory function (i.e. longterm albumin administration), decreasing the inflammatory state (i.e. statins), and reducing portal hypertension (i.e. beta-blockers).
  Arms: Comprehensive treatment

SUMMARY:
Decompensated liver cirrhosis is a life-threatening chronic liver disease with high mortality. Liver transplantation is the only option that can improve the survival of these patients; however, this procedure is associated with several limitations, such as the severe shortage of donor livers, long waiting lists, multiple complications, and high cost. Our and other previous studies have demonstrated that marrow bone-derived mesenchymal stem cells (BM-MSC) or unbilical cord derived MSC (UC-MSC) infusion is clinically safe and could improve liver function in patients with decompensated liver cirrhosis. However, the long-term outcomes of MSC infusion have not been reported until now. This prospective and randomized controlled study examined the longer-term safety and efficacy of UC-MSC in patients with decompensated liver cirrhosis.

DETAILED DESCRIPTION:
Liver cirrhosis represents a late stage of progressive hepatic fibrosis characterized by the formation and accumulation of an extracellular matrix, which leads to the progressive distortion of the hepatic architecture. In China, the most important cause of liver cirrhosis is chronic hepatitis B virus (HBV) infection. Liver cirrhosis usually progresses irreversibly into advanced stage, such as a decompensated stage which is characterized by a series of clinical manifestations, including ascites, variceal hemorrhage, and hepatic encephalopathy with high mortality. Liver transplantation is the only option that can improve the survival of these decompensated liver cirrhosis patients; however, this procedure is associated with several limitations, such as the severe shortage of donor livers, long waiting lists, multiple complications, and high cost. Therefore, it is urgent to find a safe and effective therapeutic approach to decompensated liver cirrhosis.

Animal models have shown that bone marrow-derived MSC (BM-MSC) can ameliorate liver fibrosis and reverse fulminant hepatic failure. In clinical, autologous BM-MSC have significantly improved liver function in patients with liver cirrhosis. A recent research also found that autologous BM-MSC therapy safely improved histological fibrosis and liver function in patients with alcoholic cirrhosis. Allogeneic MSC therapy, such as umbilical cord-derived MSC (UC-MSC), have shown to be safe and beneficial for the patients with liver cirrhosis caused by autoimmune diseases. Our previous studies showed that infusions of UC-MSC significantly improved liver function in decompensated liver cirrhosis and primary biliary cirrhosis (PBC) patients and increased the survival rate in acute-on-chronic liver failure (ACLF) patients. However, the single-center clinical study, the relative small size of the patient cohorts, absence of evaluation on long-term efficacy prevent firm conclusions being made with regard to the safety and efficacy of this treatment in liver diseases.

The purpose of this study is to investigate whether and how UC-MSC can improve the liver function, and the incidence of serious complications in patients with decompensated liver cirrhosis through a multi-center clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-69 years;
2. Decompensated liver cirrhosis (manifestations including gastrointestinal bleeding, hepatic encephalopathy, and ascites, based on previously stable cirrhosis);
3. Positive testing for serum hepatitis B surface antigen (HBsAg) for more than 6 months (chronic hepatitis B patients);
4. Written consent.

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies;
2. Liver cirrhosis caused by other reasons, such as autoimmune diseases, alcocal, drugs and so on;
3. Pregnant women;
4. The presence of other vital organ severe dysfunction;
5. Participate in other studies;
6. Lack of a supportive family;
7. Refusal to sign the informed consent form.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Liver function | 96 weeks
  including the levels of albumin [ALB], prothrombin activity [PTA], total bilirubin [TBIL, and cholinesterase [CHE].
The incidence of serious complications | 96 weeks
  including infection, gastrointestinal bleeding, encephalopathy, and hepatorenal syndrome.

SECONDARY OUTCOMES:
The incidence of adverse events | 96 weeks
  e.g. fever, allergy, rash, infection
Disease-free survival time | 96 weeks
  The length of survival time after first UC-MSC treatment for the patient during the follow-up period.
Incidence of hepatocellular carcinoma (HCC) events | 96 weeks
  HCC deveopled in the patient during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Study Chair — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No